CLINICAL TRIAL: NCT06114303
Title: Ex-vivo Evaluation of the Effect of 2 Probiotic Solutions (Lactibiane ATB and Lactibiane Enfant) and 5 Classes of Drugs on the Intestinal Microbiota
Acronym: EPROMED
Status: Terminated | Type: Observational
Why Stopped: This study was terminated early on 16/06/2025 because the initial results obtained from the 14 pairs of patients included were sufficient to satisfactorily address the research question posed in the context of the thesis.
Sponsor: Larena SAS (Industry)
Collaborators: Université Paris-Saclay (Other)
Responsible Party: Sponsor
Other Study IDs: PIL-RIPH3-EPROMED-023
Record Dates: First submitted 2023-02-27; First posted 2023-11-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-07

CONDITIONS: Dysbiosis
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- "Mother": Healthy women
  Interventions: Other: Stool sampling
- "Daughter": Healthy "daughter" from "Mother" subjects
  Interventions: Other: Stool sampling

INTERVENTIONS:
Other: Stool sampling — 1 stool sample is taken during the study with a stool sample kit

SUMMARY:
The objective is to test ex-vivo the effects of two probiotic solutions (Lactibiane ATB and Lactibiane Enfant) and five classes of drugs (antibiotic, proton pump inhibitor, non-steroidal anti-inflammatory, anxiolytic and anti-depressant) on microbial microcosms derived from human stool samples (from adults and children) re-cultured under anaerobic conditions.

ELIGIBILITY:
Inclusion Criteria:

Adult "Mother" population:

* Women aged 25-40 years;
* In good general health, i.e. no chronic pathology and not taking any medication at the time of inclusion and/or long-term treatment,
* With a regular bowel movement frequency (at least once every 2 days)
* BMI between 18.5 and 25
* Able and willing to participate in the research by complying with the protocol procedures
* Not objecting to the collection and processing of their personal data

Child "Daughter" population

* Girl between 1 and 2 years old
* In good general health, i.e. no chronic pathology and not taking any medication at the time of inclusion and/or on a long-term basis,
* With a regular stool frequency (at least once every 2 days)
* Whose mother does not object to the collection and processing of personal data

Exclusion Criteria:

Adult "Mother" population :

* Pregnant or breastfeeding women,
* Under antibiotic treatment, or having stopped it for less than a month.
* Under dietary supplementation (prebiotics or probiotics) or having stopped it less than one month before
* On antidepressants and/or anxiolytics in the month before inclusion
* Taking a non-steroidal anti-inflammatory drug (NSAID) the month before inclusion.
* On PPI, or having stopped it less than one month before.
* Persons under court protection,
* Person participating in another research study with an ongoing exclusion period,

Child "Daughter" population:

* Outside the WHO normal growth charts (weight for height) for girls aged 0-2 years (below the 3rd percentile or above the 97th percentile)
* Undergoing antibiotic treatment, or having stopped it less than a month ago.
* Having taken a non-steroidal anti-inflammatory drug (NSAID) in the month prior to inclusion.
* On dietary supplements (prebiotics or probiotics) or having stopped them within the last month
* Subjects participating in another research study with an ongoing exclusion period

Ages: 1 Year to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The mother/daughter " duos " participating in the study will be drawn from a panel of volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Transcriptional activity of microbiomes | 10 months
  Transcriptional activity of microbiomes by sequencing of 16S rRNA vs. the gene encoding 16S rRNA
Transcriptomic profiles of the communities | 10 months
  Transcriptomic profiles of the communities assessed by meta-transcriptomics
Metabolites produced and microbial metabolic pathways | 10 months
  Metabolites produced and microbial metabolic pathways will be assessed by global metabolomics

CONTACTS AND LOCATIONS:
Locations (1):
- Amandine FRY, Dijon, France

IPD SHARING:
Plan to Share IPD: No